CLINICAL TRIAL: NCT05699824
Title: To Study the Hemodynamic Response of Early Addition of Carvedilol to Terlipressin in Acute Variceal Bleed in Child's B and C Cirrhosis- A Randomized Controlled Trial
Brief Title: To Study the Hemodynamic Response of Early Addition of Carvedilol to Terlipressin in Acute Variceal Bleed in Child's B and C Cirrhosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-53
Record Dates: First submitted 2022-12-30; First posted 2023-01-26 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2022-12

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carvedilol at Day2 + Standard Medical Treatment (Experimental): Arm A- Carvedilol will be initiated on day 2, at a dose of 3.125mg twice a day (6.25mg/day), along with standard management as per institutional protocol for AVB.
  All patients to receive Inj. Terlipressin, 1 mg at 4 hours along with standard management for acute variceal bleed as per institutional protocol
  Interventions: Drug: Carvedilol Day2; Other: Standard Medical Treatment
- Carvedilol at Day6 + Standard Medical Treatment (Active Comparator): Arm B- Carvedilol will be initiated on day 6, at a dose of 3.125mg twice a day (6.25mg/day), along with standard management as per institutional protocol for AVB.
  All patients to receive Inj. Terlipressin, 1 mg at 4 hours along with standard management for acute variceal bleed as per institutional protocol
  Interventions: Other: Standard Medical Treatment; Drug: Carvedilol Day6

INTERVENTIONS:
Drug: Carvedilol Day2 — Carvedilol will be initiated on day 2, at a dose of 3.125mg twice a day (6.25mg/day), along with standard management as per institutional protocol for AVB.
  Arms: Carvedilol at Day2 + Standard Medical Treatment
Other: Standard Medical Treatment — All patients to receive Inj. Terlipressin, 1 mg at 4 hours along with standard management for acute variceal bleed as per institutional protocol. Standard Medical Treatment
Drug: Carvedilol Day6 — Carvedilol will be initiated on day 6, at a dose of 3.125mg twice a day (6.25mg/day), along with standard management as per institutional protocol for AVB.
  Arms: Carvedilol at Day6 + Standard Medical Treatment

SUMMARY:
Management of Acute variceal bleeding includes endoscopic variceal ligation (EVL) along with vasoactive agents. Inspite of successful hemostasis, this is associated with high variceal rebleeding (VRB) in Child B and C cirrhosis and have higher 6-week mortality rates. Pre-emptive TIPS has shown to prevent rebleed and improve survival in child B and C patients but is associated with liver related complications in advanced disease. HVPG guided therapy and treatment response is known to improve rebleeding and associated with improved survival. This is based on achieving hemodynamic response defined as HVPG reduction of ≥20% from baseline or absolute reduction of HVPG </= 12 mmHg for secondary prophylaxis for prevention of rebleeding. Studies have shown the safety of giving terlipressin in patients receiving beta- blockers. We aim to achieve hemodynamic response with addition of carvedilol with vasoactive agent for reduction of portal blood flow to decreases rebleeding episodes and reduce mortality.

DETAILED DESCRIPTION:
Aim and Objective To compare the hemodynamic response of early addition of carvedilol with terlipressin in patients with cirrhosis presenting with acute esophageal variceal bleeding.

Primary objective • To study the hemodynamic response (HVPG reduction of ≥20% from baseline or absolute reduction of HVPG </= 12 mmHg) in the groups at 5-days.

Secondary objective

* Rebleeding rate in the two groups at 5-days
* Rebleeding rate at 6-weeks
* Reduction of HVPG <16mm Hg in both groups at 5-days
* Salvage treatment, TIPS in both groups at 5-days and at 6-weeks
* Salvage treatment, SEMS, SB tube placement in-between groups at 5-days and at 6- weeks
* Survival at 6-weeks
* Liver related decompensation in-between groups at 6-weeks
* Adverse events between the groups at 6-weeks

Methodology:

Study population: Patients with Child's B and C cirrhosis who present with acute esophageal variceal bleed, between 18-75 years will be enrolled and randomized based on inclusion and exclusion criteria.

Study design- Prospective open label RCT

Study period - 1.5 years

Sample Size:Sample size will be calculated assuming that baseline characteristics (22.2±5.0 mmHg) are same and HVPG reduction on 5th day with terlipressin is 19.1±5 mmHg [7] and estimating a further reduction of 15% with addition of carvedilol [14] (16.3±4.3 mmHg), with an alpha value equal to 5 % and power of 80%, we need to enrol 45 cases in both arms. Assuming an attrition rate of 10%, it was decided to enrol 100 cases, 50 in each group, randomly allocated by block randomization method with block size of 10.

Intervention: All patients to receive Inj. Terlipressin, 1 mg at 4 hours along with standard management for acute variceal bleed as per institutional protocol

Arm A- Carvedilol will be initiated on day 2, at a dose of 3.125mg twice a day (6.25mg/day), along with standard management as per institutional protocol for AVB.

Arm B- Carvedilol will be initiated on day 6, at a dose of 3.125mg twice a day (6.25mg/day), along with standard management as per institutional protocol for AVB.

- Monitoring and assessment: Patients will be admitted in GI-bleed ICU and will be randomized into the study groups after successful endoscopic control of the bleed. Each patient will be monitored as per the institutional protocol for management of upper GI bleed. A detailed clinical history will be taken, and blood investigations and other relevant investigations required will be done as mentioned in the table 2. Patient will undergo HCC surveillance as per the guideline. Once discharged, patient will be called for OPD visits and routine investigations as planned will be done. Patient will be assessed for the tolerance of carvedilol and dose escalation to a maximum dose of 6.25mg twice a day (12.5mg/day) will be achieved. Each patient will maintain a "patient diary" for ease in recording details.

Table 2: Investigations

Day 0-5 Complete physical evaluation Hemogram, Kidney function test, Liver function test, INR Ultrasound abdomen with spleno-portal axis doppler Fibroscan-liver and spleen Coagulation parameter, vWF, ADAMTS-13 2D-ECHO, ECG Rest investigation, monitoring, antibiotics as per hospital protocol HVPG on Day 1 and at Day 5 Planned OPD visits on day 7, 14, 28, 42 Hemogram, Kidney function test, Liver function test, INR Follow-up visits Repeat upper GI endoscopy every 3 weeks till variceal eradication

Expected outcome of the project:

HVPG guided treatment and achieving hemodynamic response post bleed will reduce rebleeding rates and will prevent further decompensation and reduce mortality in patients with Child B and C cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis with Acute Variceal Bleed
* Child's B and C cirrhosis (CTP ≤ 12)
* Patients age between 18 to 75 years

Exclusion Criteria:

* Gastric variceal bleed
* Bleeding related to coagulopathy
* Other causes of portal hypertensive bleeding
* Acute on chronic liver failure
* Sepsis
* Shock(persistence of hypotension)
* Acute kidney injury (>1.5 mg%)
* Grade 3 Ascites
* Hyponatremia (Na < 125 mEq/L)
* Complete portal vein thrombosis
* Hepatocellular carcinoma (>3cm lesion)
* Tumoral portal vein thrombosis
* Chronic kidney disease
* Coronary artery disease
* Valvular heart disease
* Sick sinus syndrome/ Pacemaker
* Arrythmia
* Uncontrolled hypothyroidism and hyperthyroidism
* Pregnancy
* Failure to give consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Hemodynamic response in both groups | Day 5
  Hemodynamic response (HVPG reduction of ≥20% from baseline or absolute reduction of HVPG </= 12 mmHg) in the groups at 5-days.

SECONDARY OUTCOMES:
Rebleeding within 6-week in both groups | 6-weeks
Death in both groups | 6-weeks
Adverse Effects in both groups | 6 weeks
Decompensation events (ascites) at 6-weeks in both groups | 6 weeks
  Ascites defined as either development of ascites during the follow-up or worsening of pre-existing ascites either in the form of increasing the dose requirement of diuretic or requirement of therapeutic paracentesis.
Decompensation events (Hepatic Encephalopathy) at 6-weeks in both groups | 6 weeks
  New onset of Hepatic Encephalopathy. Hepatic encephalopathy is defined based on clinical parameters as per the West-Haven criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided